CLINICAL TRIAL: NCT01750710
Title: Correlation Between Clinical and Electrophysiological Phenotypes in a Population of Patients With Neuropathy Charcot-Marie-Tooth Disease Type 1A
Acronym: CCA1
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0128
Record Dates: First submitted 2012-11-16; First posted 2012-12-17 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Charcot-Marie-Tooth Type 1A Neuropathy
Keywords: Charcot-Marie-Tooth disease type 1A neuropathy; Isokinetic; Electromyography; Walking
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
This exploratory cross-sectional study proposes, firstly, to objectify in a population of Charcot-Marie-Tooth disease type 1A (CMT 1A)if there is a correlation between the recording of electrical parameters and upper limb muscle strength of the thigh and in a second step, to seek a relationship between the measured parameters.

DETAILED DESCRIPTION:
Patients suffering from CMT 1A neuropathy will be invited to go through a series of tests such as:

* Electromyography
* Isokinetic test
* Podiatric assessment
* Functional evaluations: Hand dexterity, limbs muscles strength
* Quality of life assessment with questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Diagnosis of Charcot Marie Tooth disease, type 1A confirmed by molecular biology (duplication 17.p11.2)
* Listening and written French
* Agreement after written information, clear and honest about the purpose of the study, the nature of the tests and their possible side effects or bothersome.
* Strength of the quadriceps superior to 2/5 MMT MRC

Exclusion Criteria:

* Presence of other neurological comorbidity
* Presence of coronary artery disease unstabilized
* Peripheral neuropathy of other causes: diabetes, monoclonal gammopathy, malignancy, solid cancer, systemic autoimmune disease (lupus, Sjögren's disease, Wegener sarcoidosis ...), infectious disease (viral hepatitis, HIV ...), drugs known to be responsible for iatrogenic neuropathy.
* Gait trouble of other origin
* Patients unable to give their consent.
* Intellectual deficit that does not allow to comply with tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from CMT 1A neuropathy
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2016-04-28 (Actual); Study Completion 2016-04-28 (Actual)

PRIMARY OUTCOMES:
axonal loss | at day 1

SECONDARY OUTCOMES:
Muscle strength | at day 1
Functional scores | at day 1
Hand testing | at day 1
spatial and temporal parameters of walking | at day 1
Barometric stabilometric podo-static scores | at day 1
Quality of life | at day 1
Fatigue | at day 1
Depression | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel COUDEYRE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Bihel L, Reynaud V, Givron P, Clavelou P, Cornut-Chauvinc C, Pereira B, Thomas E, Taithe F, Coudeyre E. Foot Function Index: A Promising Questionnaire for Individuals With Charcot-Marie-Tooth Disease Type 1A. Arch Phys Med Rehabil. 2019 Dec;100(12):2403-2406. doi: 10.1016/j.apmr.2019.06.003. Epub 2019 Jun 28. PMID 31255638